CLINICAL TRIAL: NCT04772300
Title: Prospective Multi-Center Randomized Controlled Trial to Evaluate the Safety and Efficacy of SiroLIMus Drug Coated Balloon Versus Non-coated Standard Angioplasty for the Treatment of Infrapopliteal Occlusions in Patients With PEripheral Arterial DiSease
Brief Title: Trial to Assess the Safety and Efficacy of Sirolimus-Coated Balloon vs. Uncoated Standard Angioplasty for the Treatment of Below-the-knee Peripheral Arterial Disease
Acronym: LIMES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: Concept Medical Inc. (Industry); Vascuscience (Unknown); CoreLab Black Forest (Unknown); Center for Clinical Studies Jena (Unknown)
Responsible Party: Principal Investigator, Ulf Teichgräber, Principal Coordinating Investigator, Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZKSJ0132
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Sirolimus; Drug-Coated Balloon; Percuteanous Transluminal Angioplasty; MagicTouch; Below-the-knee; BTK; Drug-Coated Ballon; plain old angioplasty; POBA; Randomized-Controlled Trial
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty

STUDY DESIGN:
Intervention Model Description: 1:1-randomization, parallel design, stratified by center.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus DCB group (Experimental): Intervention with Sirolimus-coated balloon catheter
  Interventions: Combination Product: Percutaneous Transluminal Angioplasty (PTA) MagicTouch Sirolimus Coated PTA Balloon Catheter
- POBA group (Active Comparator): Intervention with non-coated balloon catheter (POBA)
  Interventions: Device: Percutaneous Transluminal Angioplasty (PTA) with non-coated balloon catheter (POBA)

INTERVENTIONS:
Combination Product: Percutaneous Transluminal Angioplasty (PTA) MagicTouch Sirolimus Coated PTA Balloon Catheter — PTA with an sirolimus drug-coated balloon catheter (SRL-DCB) in the infrapopliteal artery
  Arms: Sirolimus DCB group
Device: Percutaneous Transluminal Angioplasty (PTA) with non-coated balloon catheter (POBA) — PTA with an non-coated balloon catheter (POBA) in the infrapopliteal artery
  Arms: POBA group

SUMMARY:
This study is a prospective, interventional, multicenter 1:1 randomized trial.

The trial evaluates the safety and efficacy of the Magic Touch PTA sirolimus drug-coated balloon in comparison to the treatment with POBA (control device) in patients with advanced infrapopliteal artery disease.

DETAILED DESCRIPTION:
The purpose of this study is to assess whether efficacy of the MagicTouch® Sirolimus Coated PTA Balloon Catheter (SRL-DCB) is superior and whether safety is non-inferior to Plain Old Balloon Angioplasty (POBA) regarding treatment of high-grade stenoses ≥ 75 % in the infrapopliteal arteries (located below the P3 segment of the popliteal artery to the tibiotalar joint) in patients presenting with chronic limb-threatening ische-mia (CLTI) (Rutherford 4-6).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of consent.
2. Subject has been informed of the nature of the study, is willing to comply with all required follow-up evaluations within the defined follow-up visit windows and has signed an Ethics Committee (EC) approved consent form.
3. Female subjects of childbearing potential have a negative pregnancy test ≤ 7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation. Female subjects will be exempted from this requirement in case they are sterile, infertile, or have been post-menopausal for at least 12 months (no menses).
4. Life expectancy > 1 year in the investigator's opinion.
5. Subject presenting with documented chronic limb-threatening ischemia (CLTI) in the target limb defined as Rutherford category 4, 5 or 6.
6. In case of Rutherford category 5 or 6: Subjects with documented infection grade ≤ 2 according to the wound ischemia foot infection (WIfI) classification.
7. All ischemia grades according to the wound ischemia foot infection (WIfI) classifi-cation are allowed.documented infection grade ≤ 2 according to the wound ischemia foot infection (WIfI) classification.

7. All ischemia grades according to the wound ischemia foot infection (WIfI) classification are allowed.

8. Reference Vessel Diameter (RVD) ≥ 2 and ≤ 4.0 mm. 9. ≥ 75 % stenosis or occlusion of the target vessel by visual estimate of the treating physician; no minimal lesion length required.

10. The target lesion may consist of multiple target vessel lesions, if they are ≤ 5 cm away from each other and if at least one of them is a stenosis ≥ 75 % and all lesions are located in only one of the infrapopliteal arteries or directly within the transition area. Non-target vessels (e.g. inflow lesions or contralateral extremity, other non-target vessels below the knee) and non-target lesions of the target ves-sel can be treated during the study index procedure but according to the patient's randomization result (interventional group: Sirolimus-coated balloon or POBA; control group: only POBA).

11. Lesion length < 30 cm, no limitation in number of used devices. 12. The lesion must be located in the infrapopliteal arteries and above the ankle joint. Lesions may not be located above the tibioperoneal trunk or below the tibiotalar joint (arteries of the foot), nor can the treatment (investigational device or standard PTA, including pre-dilatation) extend beyond these indicated regions for more than 1 cm. Note: A target lesion can extend into the P3 segment in case it involves a straight uninterrupted lesion extending from the target vessel.

13. Presence of documented run-off to the foot (clearly visible at least one of the following run-off vessels: dorsalis pedis or pedal arch or plantar arteries by angiography). The target vessel should give direct or indirect run-off to the foot.

14. Inflow free from flow-limiting lesion confirmed by angiography. Patients with flow-limiting inflow lesions (≥ 50 % stenosis) can be included if the lesion(s) have been treated successfully before enrollment, with a maximum residual stenosis of ≤ 30 % per visual assessment. If an inflow lesion must be treated within or above the P3 segment of the popliteal artery, there must be a minimum of 3 cm healthy tissue between this (treated) lesion and the infrapopliteal target lesion. Use of paclitaxel-coated devices is not permitted.

15. Successful pre-dilatation of the (entire) target lesion. Success being documented by angiographic visual estimate of ≤ 50 % residual diameter stenosis of the target lesion and no flow limiting dissection (< Grade D dissection).

16. Participants can only be enrolled once with a single target lesion.

Exclusion criteria:

1. Subjects with major amputation of the target leg above the ankle joint.
2. Planned index limb major amputation above the ankle joint, or any other planned major surgery within 30 days pre- or post-procedure. A planned amputation includ-ing and below the ankle is accepted.
3. Recent MI or stroke < 30 days prior to the index procedure.
4. Any vascular treatment with any drug-coated devices 4 weeks prior to index procedure
5. Known or suspected active infection at the time of the index procedure (abnormal white blood cell count, fever, sepsis or positive blood culture), excluding an infection of a lower extremity wound on the target limb (corresponding to WIfI infection grad 3)
6. Subjects with neurotrophic ulcers, heel pressure ulcers or calcaneal ulcers with a risk for major amputation regarding the study leg; Subjects with uncomplicated ulcers can be included.
7. Subjects with documented active osteomyelitis of the study leg, excluding the phalanges and metatarsalia, that is beyond cortical involvement of the bone per clinical judgment
8. Subjects with systemic vasculitis, such as Lupus Erythematosus or polymyalgia rheumatica on active treatment.
9. Subjects receiving systemic corticosteroid therapy (expected dosage > 5 mg of prednisolone or equivalent, per day, during the initial 9 months after procedure) or other systemic immunosuppressant therapy.
10. Known allergies or sensitivities to heparin, aspirin (ASA), other anticoagulant/antiplatelet therapies which could not be substituted, and/or sirolimus or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
11. The subject is currently enrolled in another investigational device, drug or biological trial.
12. Female subjects who are breast feeding at the time of enrollment
13. Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy
14. Prior stent(s) or bypass surgery with safety margin < 3 cm within the target vessel (including stents placed within target vessels during the index procedure prior to randomization).
15. Previous procedure with drug-coated balloons in the target vessel within 6 months prior to index procedure.
16. Stenosis ≥ 75 % or occlusions (target lesion) located or extending in the popliteal artery or below the ankle joint space. Note: A target lesion can extend into the P3 segment in case it involves a straight lesion extending from the target vessel. Non-significant stenosis below the ankle joint can be allowed in case this is not part of the target lesion.
17. Untreated significant (≥ 50 % residual stenosis measured by Duplex Sonography) inflow lesion or occlusion in the ipsilateral iliac, SFA and popliteal arteries.
18. Failure to obtain a ≤ 30 % residual stenosis in pre-existing, hemodynamically sig-nificant (≥ 50 % measured by Duplex Sonography) inflow lesions in the ipsilateral iliac, SFA and popliteal artery.
19. Aneurysm in the target vessel.
20. Angiographic evidence of thrombus within target vessel.
21. Pre-dilatation resulted in a major (≥ Grade D) flow-limiting dissection (observed on 2 orthogonal views) or residual stenosis > 50 %.
22. Use of alternative therapy, e.g. atherectomy, scoring balloon, laser, radiation therapy, stents as part of target vessel treatment or planned CO2 angiography. Note: Use of stents is only allowed for bailout stenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2028-11-17 (Estimated)

PRIMARY OUTCOMES:
composite of limb salvage and primary patency at 6 months | 6 months after study procedure (PTA with medical product under investigation or comparator)
  composite of limb salvage and primary patency at 6 months. Primary patency is defined as absence of target lesion restenosis ≥ 75 % or re-occlusion (corresponding to PSVR > 3.5 or no flow)as determined by duplex ultrasound without clinically driven target lesion revascularization (CD-TLR) after index procedure.
  Clinically driven TLR is defined as revascularization due to restenosis of ≥ 50 % in the target lesion and
  * Deterioration of Rutherford Class and/or
  * Deterioration or persistence of wounds according to the WIfI classification wound component score

SECONDARY OUTCOMES:
MALE-POD | 30 days after study procedure.
  Major Adverse Limb Events (MALE) with perioperative all-cause death (POD) at 30 days Major Adverse Limb Events (MALE) are defined as above-ankle amputation or major reintervention (i.e., new bypass graft, interposition graft revision, or thrombectomy/thrombolysis) of the treated limb involving a BTK artery.
  Perioperative death (POD) is defined as death within 30 days after index proce-dure.
  Major Adverse Limb Events (MALE) are defined as above-ankle amputation or major reintervention (i.e., new bypass graft, interposition graft revision, or thrombectomy/thrombolysis) of the treated limb involving a BTK artery.
  Perioperative death (POD) is defined as death within 30 days after index procedure.
rate of clinically-driven TVR | 1, 6, 12, 24 and 36 months after study procedure.
  occurrence of clinically-driven TVR at certain time points
TVR rate in treated target vessel and non-target vessels | 1, 6, 12, 24 and 36 months after study procedure.
  Rate of all TVR including treated non-target vessel at 1, 6, 12, 24 and 36 months.
TVR rate | 1, 6, 12, 24 and 36 months after study procedure.
  Rate of all TVR at 1, 6, 12, 24 and 36 months.
Primary Patency rate | 1, 6, 24 and 36 months after study procedure.
  Primary Patency rate at certain time points
Primary Patency of target and treat non-target vessel | 1, 6, 24 and 36 months after study procedure.
  Primary Patency rate of target and treat non-target vessel at certain time points
Secondary Patency rate | 1, 6, 24 and 36 months after study procedure.
  Secondary Patency rate at certain time points
Secondary Patency of target and treat non-target vessel | 1, 6, 24 and 36 months after study procedure.
  Secondary Patency rate of target and treat non-target vessel at certain time points
Re-stenosis of >= 75% or occlusion rate | 1, 6, 12, 24 and 36 months after study procedure.
  Rate of re-stenosis or re-occlusion at certain time points, defined as the absence of flow in the target vessel as determined by duplex ultrasound
Number of treated Non-target vessels | 36 months after study procedure
  Number of treated Non-target vessels
Walking Capacity Assessment 1 | 1, 6, 12, 24 and 36 months after study procedure.
  patient-self-assessment of walking distance at certain time points
Walking Capacity Assessment 2 | 1, 6, 12, 24 and 36 months after study procedure.
  VascuQoL questionnaire (Vascular Quality of Life Questionnaire) at certain time points; 25 questions (scale 1 to 7); best score 175, worst score 25.
Target Limb Major Amputations | 1, 6, 12, 24 and 36 months after study procedure.
  Rate of target limb major amputations at certain time points
all-cause mortality | 1, 6, 12, 24 and 36 months after study procedure.
  Rate of all-cause death at certain time points
Amputation free survival (AFS) | 1, 6, 12, 24 and 36 months after study procedure.
  Amputation free survival (AFS) at certain time points
Amputation free survival and resolved CLTI | 1, 6, 12, 24 and 36 months after study procedure.
  Amputation free survival and resolved CLTI at certain time points
Ankle-Brachial-Index (ABI) | 1, 6, 12, 24 and 36 months after study procedure.
  Change in ankle-brachial index (ABI) from pre-procedure to certain time points
Toe-Brachial-Index (TBI) | 1, 6, 12, 24 and 36 months after study procedure.
  Change in toe-brachial index (TBI) from pre-procedure to certain time points
Rutherford classification | 1, 6, 12, 24 and 36 months after study procedure.
  Change in Rutherford category from pre-procedure to certain time points
Primary sustained clinical improvement | 1, 6, 12, 24 and 36 months after study procedure.
  improvement shift in the Rutherford Category of one class or more in amputation free surviving patients without the need for clinically driven TVR at certain time points
Secondary sustained clinical improvement | 1, 6, 12, 24 and 36 months after study procedure.
  improvement shift in the Rutherford classification of one class or more in amputation free surviving patients including those with clinically driven TVR at certain time points
EQ-5D-3L | 1, 6, 12, 24 and 36 months after study procedure.
  Change in EQ-5D-3L (Quality of Life questionnaire) from pre-procedure to certain time points; 5 questions (scale 1 to 3), best score 5, worst score 15.
Wound healing | 1, 6, 12, 24 and 36 months after study procedure.
  Rate of wound healing from pre-procedure to certain time points
New or recurrent wound of the target limb | 1, 6, 12, 24 and 36 months after study procedure.
  New or recurrent wound of the target limb from pre-procedure to certain time points
Length of in-hospital-stay | 1, 6, 12, 24 and 36 months after study procedure.
  Days of hospitalization at certain time points
Major Adverse Limb Events (MALE) | 1, 6, 12, 24 and 36 months after study procedure.
  MALE at certain time points
Device Success | at index procedure
  Device Success defined as exact deployment of the device according to the instructions for use
Technical Success | at index procedure
  Technical success defined as successful vascular access and completion of the endovascular procedure with <= 50% residual diameter stenosis and restoration of in-line flow to the ankle
Procedural success | at index procedure
  30) Procedural success, defined as combination of technical success, device suc-cess and absence of major adverse events (MALE-POD, myocardial infarction, stroke) within 72 h of the index procedure).
composite endpoint: patency, rate of overall-cause death and amputation-free survival | 1, 6, 12, 24 and 36 months after study procedure.
  composite endpoint consisting of patency, rate of overall-cause death and amputation-free survival at certain time points
composite endpoint: rate of all-cause death, target limb major amputation and clinically-driven TLR | 1, 6, 12, 24 and 36 months after study procedure.
  composite endpoint consisting of rate of all-cause death, target limb major amputation and clinically-driven Target Lesion Revascularization at certain time points

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Teichgraeber, Prof. Dr., Study Director — University Hospital Jena, Institute of Radiology
Locations (19):
- Austria (2):
  - AKH Wien, Universitätsklinik für Innere Medizin II, Klinische Abteilung für Angiologie, Vienna
  - Hanusch-Krankenhaus, Vienna
- Germany (17):
  - University Hospital Tuebingen, Diagnostic and Interventional Radiology, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Hamburg-Eppendorf, Universitäres Herz- und Gefäßzentrum Hamburg, Klinik und Poliklinik für Gefäßmedizin, Hamburg, Hamburg
  - Heart and Diabetes Center North Rhine Westphalia, Clinic for General and Interventional Cardiology/Angiology, Bad Oeynhausen, North Rhine-Westphalia
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen; Clinic for Cardiology and Angiology II, Bad Krozingen
  - Universitätsklinikum Brandenburg, Abteilung für Innere Medizin 1, Hochschulklinik für Angiologie, Brandenburg
  - Sana Kliniken Oberfranken Coburg, Coburg
  - DIAKO gGmbH, Institut für Diagnostische und Interventionelle Radiologie und Neuroradiologie, Flensburg
  - Universitätsklinikum Heidelberg, Medizinische Klinik III, Kardiologie, Angiologie und Pneumologie, Heidelberg
  - Universitätsklinikum Jena, Institut für Diagnostische und Interventionelle Radiologie, Jena
  - University Hospital Leipzig, Leipzig
  - Bonifatius-Hospital Lingen (Ems), Lingen
  - Universitätsklinikum Münster, Klinik für Kardiologie I, Koronare Herzkrankheit, Herzinsuffizienz und Angiologie, Münster
  - Elblandklinikum Radebeul, Gefäßzentrum, Radebeul
  - Krankenhaus Barmherzige Brüder Regensburg, Institut für Radiologie, Neuroradiologie und Nuklearmedizin, Regensburg
  - Schön Klinik Rendsburg, Institut für Diagnostische und Interventionelle Radiologie/Neuroradiologie, Rendsburg
  - Kreiskrankenhaus Torgau, Torgau
  - GRN Klinik Weinheim, Kardiologie/Angiologie, Weinheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teichgraber U, Platzer S, Lehmann T, Ingwersen M, Aschenbach R, Beschorner U, Scheinert D, Zeller T. Sirolimus-Coated Balloon Angioplasty of Infra-popliteal Lesions for the Treatment of Chronic Limb-Threatening Ischemia: Study Protocol for the Randomized Controlled LIMES Study. Cardiovasc Intervent Radiol. 2022 Nov;45(11):1716-1724. doi: 10.1007/s00270-022-03213-z. Epub 2022 Jul 29. PMID 35906491